CLINICAL TRIAL: NCT07121140
Title: A Pilot Study of Home Blood Transfusions for Patient With Cancer Who Have Transfusion Dependent Cytopenias
Brief Title: Home Blood Transfusions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: iRISID-2024-1731; JT 44575 (Other: JeffTrial Number)
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy; Myelodysplastic Syndromes; Acute Myeloid Leukemia; Transfusion Dependent Cytopenias
Keywords: home blood transfusions; blood transfusions; RE-AIM; Supportive Care
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental - Home Blood Transfusion (Experimental): Participants will receive 1-2 blood products transfused in the home each week for a total of 5 transfusions. Participants with known RBC antibodies will only be eligible to receive platelet transfusions at home. Research nurse comes to home early to draw CBC and Type and Screen. Infusion nurse delivers blood products to home. Blood product administered. Assess vital signs following administration of blood products. Perform feasibility, acceptability, appropriateness questionnaires. Complete qualitative semi-structured interviews.
  Interventions: Procedure: Home Blood Transfusion

INTERVENTIONS:
Procedure: Home Blood Transfusion — Participants will be provided with transfusion of blood products, specifically red blood cells and platelets, in the home setting.

SUMMARY:
This is a pilot single arm study to evaluate the feasibility and acceptability of a home blood transfusion program. Patients will be enrolled with hematologic malignancies and other bone marrow failure syndromes who are transfusion dependent and interested in a home blood transfusion program. Participants enrolled in the study will receive 1-5 units of blood products at home. Data on barriers to administration will be recorded. Surveys and qualitative interviews will be completed to better understand acceptability of the program.

DETAILED DESCRIPTION:
The study is a single arm pilot study to evaluate the implementation of a novel home blood transfusion program at Thomas Jefferson University Hospital. The study population will include patients with hematologic malignancies and other bone marrow failure syndromes with transfusion dependent cytopenias. Participants will receive home blood draws and if needed same day transfusions. Data will be collected via surveys at time of each study visit, participant surveys at the end of the intervention as well as a semi structured interview. Each participant in the study will receive 1-2 blood products transfused in the home each week for a total of 5 transfusions. As a result each participant will be eligible to receive transfusions at home for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study:
* Provide signed and dated informed consent form Willing to comply with all study procedures and be available for the duration of the study
* Male or female, over the age of 18
* Must meet definition of transfusion dependence (require at least 2 blood product transfusions over a 28-day period)
* Receive their cancer care at SKCCC
* Have a history of blood product transfusions and NO history of transfusion reactions,
* Live within a 30-mile range of the Center City SKCCC location.
* Must be willing to allow people into the home

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:
* Patients who have a history of a transfusion reaction
* Heart failure as defined by AHA stage C or NYHA Class II-IV
* Non-English or Spanish speaking
* Are unhoused
* Are incarcerated
* Have poor venous access
* Diagnosis of Solid Tumor malignancy
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a home blood transfusion program utilizing the RE-AIM framework | 5 weeks
  The feasibility of the program defined as greater than 80% of home blood product transfusions occur as planned.
Acceptability of a home blood transfusion program utilizing the RE-AIM framework | 5 weeks
  Surveys and qualitative interviews will be completed to better understand acceptability of the program. Acceptability will be measured using the acceptability of intervention measure.
  Based on a 5-point Likert scale. Score range: 1 (Completely Disagree) to 5 (Completely Agree)

SECONDARY OUTCOMES:
Evaluate patient perspective of home blood transfusions via qualitative analysis. | Within 3 weeks of final home transfusion
  Evaluate patient perspective of home blood transfusions via qualitative analysis. Semi-structured interviews will be evaluated through qualitative analysis. All interviews will be digitally recorded and transcribed. Interviews will be analyzed using NVIVO software for coding and analysis. The codebook will be developed using conventional content analysis. All members of the research team will read the first three transcripts and identify concepts, leading to the initial code structure. This initial code structure will be applied to subsequent interviews by two coders and refined to include new themes as they emerge. This iterative process will continue until coders and at least one other team member agree upon a final coding structure, with discrepancies resolved through consensus. The two coders will apply the final structure to all transcripts. Coders will double code about 30-40% of the transcripts. Intercoder reliability will be calculated in NVivo 12 using the κ coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Binder, MD, Principal Investigator — Adam.Binder@jefferson.edu
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Vijenthira A, Starkman R, Lin Y, Stanworth SJ, Bowen D, Harrison L, Wintrich S, Callum J, Buckstein R. Multi-national survey of transfusion experiences and preferences of patients with myelodysplastic syndrome. Transfusion. 2022 Jul;62(7):1355-1364. doi: 10.1111/trf.16946. Epub 2022 Jun 10. PMID 35686926
- [Background] Garcia D, Aguilera A, Antolin F, Arroyo JL, Lozano M, Sanroma P, Romon I. Home transfusion: three decades of practice at a tertiary care hospital. Transfusion. 2018 Oct;58(10):2309-2319. doi: 10.1111/trf.14816. Epub 2018 Sep 19. PMID 30229938
- [Background] Niscola P, Tendas A, Giovannini M, Cupelli L, Trawinska MM, Palombi M, Scaramucci L, Brunetti GA, Perrotti A, Neri B, Efficace F, Cartoni C, de Fabritiis P, Mandelli F. Transfusions at home in patients with myelodysplastic syndromes. Leuk Res. 2012 Jun;36(6):684-8. doi: 10.1016/j.leukres.2012.01.010. Epub 2012 Feb 14. PMID 22336393
- [Background] Charron J, Gouezec H, Bajeux E. [Home blood transfusion in France: Benefits and development terms]. Transfus Clin Biol. 2019 Nov;26(4):304-308. doi: 10.1016/j.tracli.2018.08.161. Epub 2018 Sep 12. French. PMID 30268597
- [Background] LeBlanc TW, Egan PC, Olszewski AJ. Transfusion dependence, use of hospice services, and quality of end-of-life care in leukemia. Blood. 2018 Aug 16;132(7):717-726. doi: 10.1182/blood-2018-03-842575. Epub 2018 May 30. PMID 29848484
- [Background] Odejide OO, Steensma DP. Patients with haematological malignancies should not have to choose between transfusions and hospice care. Lancet Haematol. 2020 May;7(5):e418-e424. doi: 10.1016/S2352-3026(20)30042-9. PMID 32359453
- [Background] Thompson HW, McKelvey J. Home blood transfusion therapy: a home health agency's 5-year experience. Transfusion. 1995 May;35(5):453. doi: 10.1046/j.1537-2995.1995.35595259158.x. No abstract available. PMID 7740619
- [Background] Koepke MD, Nyman JA, Koepke JA. Home blood transfusions: the medical, economic, and legal issues surrounding a new treatment procedure. J Health Polit Policy Law. 1988 Fall;13(3):565-79. doi: 10.1215/03616878-13-3-565. PMID 3049774
- [Background] Benson K, Popovsky MA, Hines D, Hume H, Oberman HA, Glassman AB, Pisciotto PT, Thurer RL, Stehling L, Anderson KC. Nationwide survey of home transfusion practices. Transfusion. 1998 Jan;38(1):90-6. doi: 10.1046/j.1537-2995.1998.38198141505.x. PMID 9482401
- [Background] de Swart L, Smith A, Johnston TW, Haase D, Droste J, Fenaux P, Symeonidis A, Sanz G, Hellstrom-Lindberg E, Cermak J, Germing U, Stauder R, Georgescu O, MacKenzie M, Malcovati L, Holm MS, Almeida AM, Madry K, Slama B, Guerci-Bresler A, Sanhes L, Beyne-Rauzy O, Luno E, Bowen D, de Witte T. Validation of the revised international prognostic scoring system (IPSS-R) in patients with lower-risk myelodysplastic syndromes: a report from the prospective European LeukaemiaNet MDS (EUMDS) registry. Br J Haematol. 2015 Aug;170(3):372-83. doi: 10.1111/bjh.13450. Epub 2015 Apr 24. PMID 25907546
- [Background] Cannas G, Fattoum J, Raba M, Dolange H, Barday G, Francois M, Elhamri M, Salles G, Thomas X. Transfusion dependency at diagnosis and transfusion intensity during initial chemotherapy are associated with poorer outcomes in adult acute myeloid leukemia. Ann Hematol. 2015 Nov;94(11):1797-806. doi: 10.1007/s00277-015-2456-2. Epub 2015 Jul 23. PMID 26202609
- [Background] Jiang C, Yabroff KR, Deng L, Wang Q, Perimbeti S, Shapiro CL, Han X. Self-reported Transportation Barriers to Health Care Among US Cancer Survivors. JAMA Oncol. 2022 May 1;8(5):775-778. doi: 10.1001/jamaoncol.2022.0143. PMID 35323841
- [Background] Doshi R, Gonzalez KM, Hossain A, Gentsch AT, Vivero A, Wilde L, Rising KL, Binder AF. MD Perceptions of a home blood transfusion program among patients with hematologic malignancies who are newly diagnosed as compared to those with relapsed/refractory disease American Society of Hematology Conference 2023
- [Background] Andersen SK, Croxford R, Earle CC, Singh S, Cheung MC. Days at Home in the Last 6 Months of Life: A Patient-Determined Quality Indicator for Cancer Care. J Oncol Pract. 2019 Apr;15(4):e308-e315. doi: 10.1200/JOP.18.00338. Epub 2019 Mar 8. PMID 30849006
- [Background] Banerjee R, George M, Gupta A. Maximizing Home Time for Persons With Cancer. JCO Oncol Pract. 2021 Sep;17(9):513-516. doi: 10.1200/OP.20.01071. Epub 2021 Mar 4. No abstract available. PMID 33661703
- [Background] Saleem R, MacDougall K, Hassan A, et al. Novel Home-Based Transfusion Model of Palliative Care in Malignant Hematology. Blood (2022) 140 (Supplement 1): 11024- 11025.
- [Background] Craig JI, Milligan P, Cairns J, McClelland DB, Parker AC. Nurse practitioner support for transfusion in patients with haematological disorders in hospital and at home. Transfus Med. 1999 Mar;9(1):31-6. doi: 10.1046/j.1365-3148.1999.009001031.x. PMID 10216903
- [Background] Barki-Harrington L, Baron-Epel O, Shaulov A, Akria L, Barshay Y, Dally N, Deshet D, Inbar T, Koren-Michowitz M, Leiba M, Moshe Y, Shvidel L, Tadmor T, Yagenah S, Zektser M, Preis M, Hellman I, Yahalom V, Aviv A. Willingness and concerns of transfusion-dependent hematological patients toward the option of home transfusion therapy. Palliat Med. 2021 May;35(5):927-932. doi: 10.1177/02692163211000634. Epub 2021 Mar 24. PMID 33761783
- [Background] Athilingam P, D'aoust R, Zambroski C, et al. Predictive Validity of NYHA and ACC/AHA Classifications of Physical and Cognitive Functioning in Heart Failure, International Journal of Nursing Science, Vol. 3 No. 1, 2013, pp. 22-32. doi: 10.5923/j.nursing.20130301.04.
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Viera AJ, Garrett JM. Understanding interobserver agreement: the kappa statistic. Fam Med. 2005 May;37(5):360-3. PMID 15883903
- [Background] Yao R, Zhang W, Evans R, Cao G, Rui T, Shen L. Inequities in Health Care Services Caused by the Adoption of Digital Health Technologies: Scoping Review. J Med Internet Res. 2022 Mar 21;24(3):e34144. doi: 10.2196/34144. PMID 35311682